CLINICAL TRIAL: NCT03607227
Title: Does Continuous Popliteal Nerve Block Improve Pain Management for Patients Undergoing Major Maxilla or Mandible Resection With Microvascular Reconstruction Using a Free Fibula Graft
Brief Title: Continous Popliteal Block for Microvascular Free Flap Reconstruction in Ear, Nose and Throat Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Region Skane 20180602
Record Dates: First submitted 2018-06-20; First posted 2018-07-31 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Cancer; Pain, Musculoskeletal
Keywords: microsurgical free flaps; popliteal nerve block; head and neck cancer; postoperative pain
MeSH Terms: conditions — Head and Neck Neoplasms; Musculoskeletal Pain; Pain, Postoperative | interventions — Levobupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local anesthetic (Active Comparator): Levobupivacaine 3.75 mg/ml 15 ml is given as a bolus injection at start of surgery, followed by ropivacaine 2 mg/ml continous infusion 5-8 ml/h from the end of surgery until end of intervention at the fourth to seventh postoperative day.
  Interventions: Drug: Levobupivacaine
- Saline (Placebo Comparator): Saline solution (NaCl 0.9%) is given in equivalent intervals and doses as in the active substance arm.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Levobupivacaine — Active substance. Levobupivacaine 3.75 mg/ml 15 ml is given as a bolus injection at start of surgery, followed by ropivacaine 2 mg/ml continous infusion 5-8 ml/h from the end of surgery until end of intervention at the fourth to seventh postoperative day.
  Arms: Local anesthetic
Drug: Saline Solution — Placebo. Saline solution (NaCl 0.9%) is given in equivalent intervals and doses as the active substances.
  Arms: Saline

SUMMARY:
The aim of the study is to assess the effects of a continuous popliteal block on postoperative pain and recovery after major ear, nose and throat surgery with microvascular free flap reconstruction using a fibula graft.

DETAILED DESCRIPTION:
Tumors of the head and neck is one of the most common cancer types, and the incidence is increasing. Management of these tumors is complex, and treatment can include surgery with extensive resection of the mandible or maxilla, which requires reconstruction using a microvascular free flap, oftentimes a part of the fibula. The injury to the operated leg can cause significant postoperative pain, which in these patients traditionally has been treated with intravenous opioids. These drugs have good analgesic properties, but also several side effects, such as fatigue, nausea and respiratory depression. The experience at Skåne University hospital in Lund has also been that the analgesic effect in the leg has been insufficient. The investigators would therefore like to evaluate the effect of adding a continuous popliteal block on postoperative pain and opioid consumption, as well as postoperative recovery. This type of block is regularly used for orthopedic surgery of the fibula, but its effects and significance have not been evaluated for the patient group in question.

Patients will receive information about the study and, if they opt to participate, be included during the routine preoperative visit. All patients included in the study will preoperatively receive a popliteal nerve block catheter in technical accordance with local procedure guidelines, and be randomized to either active substance (local anesthetic) or placebo (saline solution). They will receive a bolus injection of the allotted substance (blinded to both patient, care provider and investigator) at the start of surgery, followed by continuous infusion during the first, maximally, seven days. During this period pain, nausea and vomiting, as well as sensory and motor function in the operated leg will be recorded regularly. Opioid consumption, need for other analgesics and ability to mobilize will also be noted. Follow up of above mentioned parameters will be made at the first routine office visit at three months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Skåne University hospital department of ear, nose and throat surgery undergoing major resection of maxilla or mandible and reconstruction using free fibula graft.
* Preoperatively able to walk (with or without aid).

Exclusion Criteria:

* Neurological disease or peripheral neuropathy affecting the donor leg of the fibula graft.
* Conditions of coagulopathy, or treatment with anticoagulant drugs, that contraindicates peripheral nerve block according to local guidelines.
* Local anesthetic allergy.
* Inability to understand study information or answer questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessed by VAS (ranging from 0 (no pain) to 10 (worst possible pain)). | Assessment of pain using VAS three times a day during the first seven postoperative days, with follow-up at the first office visit three months after surgery.
  Change in pain in the operated leg, measured with visual analogue scale (VAS), between the two study groups (the two study arms described above). VAS assesses self-perceived pain. The scale ranges from 0 (meaning no pain at all) to 10 (meaning worst possible pain). Low VAS scores (representing no to low pain) are better than high VAS scores (representing severe pain).

SECONDARY OUTCOMES:
Postoperative nausea, assessed by VAS (ranging from 0 (no nausea) to 10 (worst possible nausea)), and vomiting (yes/no). | Assessment of nausea using VAS and occurence of vomiting (yes/no) three times a day during the first seven postoperative days, with follow-up assessment of nausea at the first office visit three months after surgery.
  Change in nausea, measured with visual analogue scale (VAS), and occurence of vomiting (yes/no), between the two study groups (the two study arms described above). VAS assesses self-perceived nausea. The scale ranges from 0 (meaning no nausea at all) to 10 (meaning worst possible nausea). Low VAS scores (representing none to little nausea) are better than high VAS scores (representing severe nausea).
Postoperative sensory and motor function in the operated leg assessed by a simplified scale (ranging from 0 to 2, see description below). | Assessment of sensory and motor function using the scale described above three times a day during the first seven postoperative days, with follow-up assessment at the first office visit three months after surgery.
  Change in sensory and motor function in the operated leg between the two study groups (the two study arms described above) is assessed using a local simplified scale. The intervals are 0 (meaning no impact on sensory/motor function), 1 (meaning some impact on sensory/motor function) and 2 meaning severe impact on sensory/motor) function. Sensory function is self-perceived during touching of the forefoot, while motor function (tested as flexion of the ankle and toes) is evaluated by the investigator. Low scores (representing no or little impact on sensory/motor function) are better than high scores (indicating more impact on sensory/motor function).
Ability of postoperative mobilization (sitting/standing/walking, with or without tools/aids). | Assessment of level of mobilization (sitting/standing/walking) three times a day during the first seven postoperative days, with follow-up assessment at the first office visit three months after surgery.
  Ability of/level of postoperative mobilization (sitting/standing/walking). Tools/aids (walker/cain/staff members) needed are reported (if any).
Opioid consumption in the postoperative period. | Notation of the amount of opioids (preparation, route and dose) consumed is noted daily during the first seven postoperative days, with follow-up assessment at the first office visit three months after surgery.
  Amount of opioids needed in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Walther Sturesson, MD, PhD, Principal Investigator — Skåne University hospital, Region Skåne
Locations (1):
- Skane University Hospital Lund, Divison of Anaestesia and Intensive Care, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marur S, Forastiere AA. Head and Neck Squamous Cell Carcinoma: Update on Epidemiology, Diagnosis, and Treatment. Mayo Clin Proc. 2016 Mar;91(3):386-96. doi: 10.1016/j.mayocp.2015.12.017. PMID 26944243
- [Background] Ragbir M, Brown JS, Mehanna H. Reconstructive considerations in head and neck surgical oncology: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S191-S197. doi: 10.1017/S0022215116000621. PMID 27841135
- [Background] Dort JC, Farwell DG, Findlay M, Huber GF, Kerr P, Shea-Budgell MA, Simon C, Uppington J, Zygun D, Ljungqvist O, Harris J. Optimal Perioperative Care in Major Head and Neck Cancer Surgery With Free Flap Reconstruction: A Consensus Review and Recommendations From the Enhanced Recovery After Surgery Society. JAMA Otolaryngol Head Neck Surg. 2017 Mar 1;143(3):292-303. doi: 10.1001/jamaoto.2016.2981. PMID 27737447
- [Background] Borgeat A, Blumenthal S, Lambert M, Theodorou P, Vienne P. The feasibility and complications of the continuous popliteal nerve block: a 1001-case survey. Anesth Analg. 2006 Jul;103(1):229-33, table of contents. doi: 10.1213/01.ane.0000221462.87951.8d. PMID 16790658
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643